CLINICAL TRIAL: NCT04593472
Title: Sharing Healthcare Wishes in Primary Care
Brief Title: SHARE: Sharing Healthcare Wishes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MedStar Health (Other); Johns Hopkins Community Physicians (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB00242431; R01AG058671 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Impairment
Keywords: Cognitive Impairment; Primary Care
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHARE (Experimental): SHARE components include: 1) a letter from the practice introducing the initiative, 2) access to a designated person (medical assistant, social worker, nurse, or lay person) trained to lead advance care planning discussions, 3) person-family agenda-setting to align perspectives about the role of the caregiver and stimulate discussion about goals of care, and 4) education about communication and available resources, including a 44-page brochure developed by the National Institute on Aging entitled "A Guide for Older People: Talking with your Doctor", a blank easy to complete advance directive, and facilitated registration to the patient portal (for patient and caregiver participants) to extend electronic interactions and information access to family.
  Interventions: Behavioral: Sharing Healthcare Wishes in Primary Care (SHARE)
- Minimally Enhanced Usual Care (Placebo Comparator): Minimally enhanced usual care participants are provided with print educational materials that include a 44-page brochure developed by the National Institute on Aging entitled "A Guide for Older People: Talking with your Doctor" and a blank easy-to-complete advance directive.
  Interventions: Behavioral: Minimally Enhanced Usual Care

INTERVENTIONS:
Behavioral: Sharing Healthcare Wishes in Primary Care (SHARE) — SHARE is a multicomponent communication intervention to proactively engage family members or friends to support advance care planning in primary care.
  Arms: SHARE
Behavioral: Minimally Enhanced Usual Care — Minimally enhanced usual care participants are provided with print educational materials that include a 44-page brochure developed by the National Institute on Aging entitled "A Guide for Older People: Talking with your Doctor" and a blank easy-to-complete advance directive.
  Arms: Minimally Enhanced Usual Care

SUMMARY:
This study evaluates the efficacy of Sharing Healthcare Wishes in Primary Care (SHARE), a two-group randomized trial at up to 9 primary care practices in which 124 dyads receive a control protocol of minimally enhanced usual care and 124 dyads receive the SHARE protocol. This study tests the efficacy of SHARE on quality of communication (primary outcome) and advance care planning processes (secondary outcomes) at 6 months among primary care patients with cognitive impairment (mild-severe) and family caregiver dyads. For patients who die while enrolled in the study by 24 months, this study examines the quality of end-of-life care and bereaved family caregiver experiences with medical decision-making (secondary outcomes).

DETAILED DESCRIPTION:
SHARE is guided by the patient-provider communication, family caregiving, health services, and health informatics literatures in acknowledging the multiple pathways by which interpersonal relationships influence treatment decisions and end-of-life care. Each component of SHARE has been found to improve a range of communication outcomes in other care contexts, but have not previously been applied in this combination or examined with regard to advance care planning in persons with cognitive impairment. SHARE is designed to be broadly scalable and widely relevant to diverse primary care patients and stakeholders. The study goal is to engage family members or friends ("family" and/or "caregiver") in longitudinal interactions with primary care clinicians and stimulate and support advance care planning discussions in primary care. SHARE seeks to improve communication for persons with cognitive impairment by establishing a structured protocol to proactively engage family caregivers in ongoing interactions with primary care clinicians and stimulate and support advance care planning in primary care throughout the disease trajectory.

SHARE evaluates a multicomponent communication intervention to proactively engage family members or friends and support advance care planning in primary care. SHARE encompasses the following four therapeutic elements: 1) a letter from the practice introducing the initiative, 2) access to a designated person (medical assistant, social worker, nurse, or lay person) trained to lead advance care planning discussions, 3) person-family agenda-setting to align perspectives about the role of the caregiver and stimulate discussion about goals of care, and 4) education about communication and available resources, including a 44-page brochure developed by the National Institute on Aging entitled "A Guide for Older People: Talking with your Doctor", a blank easy to complete advance directive, and facilitated registration to the patient portal (for patient and caregiver) to extend electronic interactions and information access to family. The control group receives minimally enhanced usual care with print educational materials that include the 44-page brochure developed by the National Institute on Aging entitled "A Guide for Older People: Talking with your Doctor" and a blank easy-to-complete advance directive. Participants in both groups are followed over a 24-month period. Outcomes are assessed from patient and caregiver enrollment surveys conducted in-person or by telephone or video conference at enrollment and follow-up telephone or web surveys at 6, 12, and 24 months; Electronic health record portal activity; information about advance directive completion from the electronic medical record; burdensome care at the end of life from family survey and Chesapeake Regional Information System for our Patients (CRISP).

ELIGIBILITY:
Inclusion Criteria:

* Patient: 80 years or older, English speaking, able to provide informed consent themselves or through their legally authorized representative, identify a family member or friend who plays an active role in care coordination or accompanies them to primary care visits, not planning to move out of state within the next year, and cognitive impairment (mild-severe) on the basis of one or more incorrect answers or not being able to respond to a validated 6-item telephone screening instrument.
* Family/Friend: 18 years and older, English speaking, hear well enough to communicate by telephone, not planning to move out of the state within the next year, do not report having a life-threatening illness and are a family member or unpaid friend who attends at least some medical visits of an eligible person with cognitive impairment, do not screen positive as having cognitive impairment on the basis of fewer than two incorrect answers on the 6-item telephone screening instrument.

Exclusion Criteria:

* Patient: less than 80 years old, non-English speaking, do not help with care coordination or attend primary care visits with a family member/friend, no willing/able legal guardian or representative to provide written informed consent for those who do not have capacity, plan to move out of state within the next year, or do not have cognitive impairment on the basis of all correct answers on the 6-item telephone screening instrument.
* Family/Friend: less than 18 years old, non-English speaking, do not help with care coordination or attend at least some medical visits of an eligible patient, do not hear well enough to communicate by telephone, report having a life-threatening illness, plan to move out of state within the next year, are a non-family member who is paid for their services, or has cognitive impairment on the basis of two or more incorrect answers on the 6-item telephone screening instrument.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 273 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wolff, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (9):
- United States (9):
  - Johns Hopkins Community Physicians - Remington, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Beacham Center, Baltimore, Maryland
  - Medstar Harbor Hospital, Baltimore, Maryland
  - Johns Hopkins Community Physicians - Greater Dundalk, Dundalk, Maryland
  - Medstar CSA Collington and House call Program, Mitchellville, Maryland
  - Johns Hopkins Community Physicians - White Marsh, Nottingham, Maryland
  - Medstar CSA Montgomery County, Olney, Maryland
  - MedStar Health at Leisure World Boulevard, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff JL, Berger A, Clarke D, Green JA, Stametz R, Yule C, Darer JD. Patients, care partners, and shared access to the patient portal: online practices at an integrated health system. J Am Med Inform Assoc. 2016 Nov;23(6):1150-1158. doi: 10.1093/jamia/ocw025. Epub 2016 Mar 28. PMID 27026614
- [Background] Wolff JL, Aufill J, Echavarria D, Heughan JA, Lee KT, Connolly RM, Fetting JH, Jelovac D, Papathakis K, Riley C, Stearns V, Thorner E, Zafman N, Levy HP, Dy SM, Wolff AC. Sharing in care: engaging care partners in the care and communication of breast cancer patients. Breast Cancer Res Treat. 2019 Aug;177(1):127-136. doi: 10.1007/s10549-019-05306-9. Epub 2019 Jun 4. PMID 31165374
- [Background] Wolff JL, Roter DL, Boyd CM, Roth DL, Echavarria DM, Aufill J, Vick JB, Gitlin LN. Patient-Family Agenda Setting for Primary Care Patients with Cognitive Impairment: the SAME Page Trial. J Gen Intern Med. 2018 Sep;33(9):1478-1486. doi: 10.1007/s11606-018-4563-y. Epub 2018 Jul 18. PMID 30022409
- [Background] Wolff JL, Cagle J, Echavarria D, Dy SM, Giovannetti ER, Boyd CM, Hanna V, Hussain N, Reiff JS, Scerpella D, Zhang T, Roth DL. Sharing Health Care Wishes in Primary Care (SHARE) among older adults with possible cognitive impairment in primary care: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Jun;129:107208. doi: 10.1016/j.cct.2023.107208. Epub 2023 Apr 26. PMID 37116645
- [Background] Cagle JG, Reiff JS, Smith A, Echavarria D, Scerpella D, Zhang T, Roth DL, Hanna V, Boyd CM, Hussain NA, Wolff JL. Assessing Advance Care Planning Fidelity within the Context of Cognitive Impairment: The SHARE Trial. J Pain Symptom Manage. 2024 Aug;68(2):180-189. doi: 10.1016/j.jpainsymman.2024.05.002. Epub 2024 May 15. PMID 38754769
- [Background] Wolff JL, Cagle JG, Hanna V, Dy SM, Echavarria D, Giovannetti ER, Boyd CM, Saylor MA, Hussain N, Reiff JS, Scerpella D, Zhang T, Sekhon VK, Roth DL. Sharing health care wishes among older adults with cognitive impairment in primary care: Results from a randomized controlled trial. Alzheimers Dement. 2024 Oct;20(10):7263-7273. doi: 10.1002/alz.14210. Epub 2024 Aug 27. PMID 39189632
- [Derived] Reiff JS, Cagle J, Zhang T, Roth DL, Wolff JL. Fielding the quality of communication questionnaire to persons with cognitive impairment and their family in primary care: A pilot study. J Am Geriatr Soc. 2023 Jan;71(1):221-226. doi: 10.1111/jgs.18034. Epub 2022 Sep 6. PMID 36069000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 primary care practices at two health systems from October 2020 to December 2022. Both patient and care partner must have been eligible to participate. Eligible patients were ≥80 years and screened positive for cognitive impairment (1+ incorrect answer or unable to respond to a 6-item screening survey). Eligible care partners were ≥18 years, English-speaking, no life-threatening illness, and did not screen positive for cognitive impairment.
Pre-assignment Details: Of 4,441 patient-family dyads who were outreached, 606 opted out of the study via opt-out card, and 3,835 were screened. Of 3,835 screened, 3,557 were ineligible (369 unreachable, 2,458 did not meet eligibility criteria, 730 refused, 5 consented not randomized due to lost to follow up). Patient and caregivers were enrolled as dyads. A total of 273 patient-family dyads were enrolled and randomized. The total number of individual participants is 546 (Participants started in Protocol Section).
Groups:
- SHARE Group: Of 273 enrolled patient-family dyads, 145 were randomized to the SHARE intervention group and received a packet from the primary care practice including a person-family agenda setting checklist, blank advance directive, guide for communication with clinicians, instructions for completing proxy registration for the patient portal and an invitation to a facilitator led advance care planning (ACP) conversation.
- Control Group: Of 273 enrolled patient-family dyads, 128 were assigned to the control group and received minimally enhanced usual care encompassing an introductory letter, the guide for communicating with clinicians and blank advance directive.
Period: Overall Study
Arm/Group | SHARE Group | Control Group
Started | 145 (145 patients and 145 caregivers started the study in the intervention group The total number of individual participants who started the study in the intervention group is 290.) | 128 (128 patients and 128 caregivers started the study in the control group. The total number of individual participants who started the study in the control group is 256.)
Completed 6-Month Follow-Up Interview | 108 (108 patients and 108 caregivers completed the 6-month milestone in the intervention group. The total number of individual participants who completed the 6-month milestone in the intervention group is 216.) | 97 (97 patients and 97 caregivers completed the 6-month milestone in the control group. The total number of individual participants who completed the 6-month milestone in the control group is 194.)
Completed 12-Month Follow-Up Interview | 86 (86 patients and 86 caregivers completed the 12-month milestone in the intervention group. The total number of individual participants who completed the 12-month milestone in the intervention group is 172.) | 77 (77 patients and 77 caregivers completed the 12-month milestone in the control group. The total number of individual participants who completed the 12-month milestone in the control group is 154.)
Completed | 47 (47 patients and 47 caregivers completed the 24-month milestone in the intervention group. The total number of individual participants who completed the 24-month milestone in the intervention group is 94.) | 49 (49 patients and 49 caregivers completed the 24-month milestone in the control group. The total number of individual participants who completed the 24-month milestone in the control group is 98.)
Not Completed | 98 | 79
Not completed — Death | 31 | 27
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Dropped due to provider change between either 6, 12 or 24 months | 33 | 22
Not completed — Dropped due to caregiver change between either 6, 12 or 24 months | 5 | 4
Not completed — Dropped due to participants missing assessment at both 6 and 12-month | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Still collecting 24-month assessment | 17 | 10

BASELINE CHARACTERISTICS:
Population: Patients and Caregivers
Groups:
- SHARE Group: Of 273 patient-family dyads enrolled, 145 patients and 145 caregivers were randomized to the SHARE intervention group and received a packet from the primary care practice including a person-family agenda setting checklist, blank advance directive, guide for communication with clinicians, instructions for completing proxy registration for the patient portal and an invitation to a facilitator led ACP conversation. A total of 290 participants were randomized to the SHARE intervention group.
- Control Group: Of 273 patient-family dyads enrolled, 128 patients and 128 caregivers were assigned to the control group and received minimally enhanced usual care encompassing an introductory letter, the guide for communicating with clinicians and blank advance directive. A total of 256 participants were randomized to the control group.
- Total: Total of all reporting groups
Arm/Group | SHARE Group | Control Group | Total
Number analyzed (Participants) | 290 | 256 | 546
Age, Categorical [Count of Participants; unit: Participants] — Population: The row population for each row (patient and caregiver) differs from the overall number of baseline participants because each row specifies the number of participants analyzed separately by patient or caregiver.
  Participants
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient: <=18 years | 0 | 0 | 0
    Patient: Between 18 and 65 years | 0 | 0 | 0
    Patient: >=65 years | 145 | 128 | 273
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver: <=18 years | 0 | 0 | 0
    Caregiver: Between 18 and 65 years | 81 | 67 | 148
    Caregiver: >=65 years | 64 | 61 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The row population for each row (patient and caregiver) differs from the overall number of baseline participants because each row specifies the number of participants analyzed separately by patient or caregiver.
  years
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient | 88.0 (5.9) | 87.9 (5.8) | 88.0 (5.8)
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver | 65.7 (10.8) | 66.3 (13.6) | 66.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The row population for each row (patient and caregiver) differs from the overall number of baseline participants because each row specifies the number of participants analyzed separately by patient or caregiver.
  Participants
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient: Female | 89 | 82 | 171
    Patient: Male | 56 | 46 | 102
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver: Female | 122 | 101 | 223
    Caregiver: Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The row population for each row (patient and caregiver) differs from the overall number of baseline participants because each row specifies the number of participants analyzed separately by patient or caregiver.
  Participants
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient: Hispanic or Latino | 6 | 3 | 9
    Patient: Not Hispanic or Latino | 139 | 125 | 264
    Patient: Unknown or Not Reported | 0 | 0 | 0
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver: Hispanic or Latino | 6 | 4 | 10
    Caregiver: Not Hispanic or Latino | 139 | 122 | 261
    Caregiver: Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The row population for each row (patient and caregiver) differs from the overall number of baseline participants because each row specifies the number of participants analyzed separately by patient or caregiver.
  Participants
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient: Black | 46 | 30 | 76
    Patient: Asian | 6 | 7 | 13
    Patient: White | 88 | 86 | 174
    Patient: Other race/missing | 5 | 5 | 10
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver: Black | 45 | 31 | 76
    Caregiver: Asian | 5 | 5 | 10
    Caregiver: White | 90 | 84 | 174
    Caregiver: Other race/missing | 5 | 8 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 290 | 256 | 546
Education >12th grade [Count of Participants; unit: Participants] — Population: Patients' and Caregivers' measures were assessed separately.
  Participants
    Patient: number analyzed (Participants) | 145 | 128 | 273
    Patient | 72 | 69 | 141
    Caregiver: number analyzed (Participants) | 145 | 128 | 273
    Caregiver | 121 | 96 | 217
Patient Diagnosis of Cognitive Impairment [Count of Participants; unit: Participants] — Population: Patients only
  Participants
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 71 | 63 | 134
Patient - Moderate or Severe Cognitive Impairment (based on TICS-m score) [Count of Participants; unit: Participants] — We use the Modified Telephone Interview for Cognitive Status (TICS-m) to categorize normal cognitive functioning (scores of 32-50), mild cognitive impairment (scores of 28-31) or severe (scores of less than 27) cognitive impairment. Population: Patients only.
  Participants
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 108 | 81 | 189
Patient - Live Alone [Count of Participants; unit: Participants] — Population: Patient only
  Participants
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 40 | 41 | 81
Caregiver Relationship to Patient [Count of Participants; unit: Participants] — This measure was only assessed for the caregivers. Population: The row population differs from the overall number of participants because this measure was only assessed for the caregiver population.
  Participants
    number analyzed (Participants) | 145 | 128 | 273
    Spouse/Partner | 33 | 36 | 69
    Adult Child | 103 | 82 | 185
    Other (friend, other relative) | 9 | 10 | 19
Patient Reported Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Quality of Life Alzheimer's Disease (QoL-AD) scale is dementia specific and brief and uses the patient's own responses. It has 13 items covering the domains of physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole. These are scored on a 4-point Likert scale, ranging from 1 (poor) to 4 (excellent), with a possible total range from 13 to 52. Higher scores indicate better quality of life. Population: Patient only
  score on a scale
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 34.5 (7.0) | 35.4 (6.5) | 34.9 (6.8)
Caregiver Reported Fair or Poor Self-rated Health [Count of Participants; unit: Participants] — Caregivers were asked to rate their physical health using a 4-item Likert scale (poor, fair, good or excellent). The number of caregivers indicating poor or fair physical health is reported. Population: Caregivers only
  Participants
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 22 | 17 | 39
Caregiver Reported - Hours helping patient in a typical week [Mean (Standard Deviation); unit: hours/week] — Caregivers were asked to estimate the number of hours in a typical week spent helping the enrolled patient. Population: Caregivers only
  hours/week
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 25.7 (33.3) | 22.4 (32.7) | 24.1 (33.0)
Caregiver Reported - Years accompanying patients to visits [Mean (Standard Deviation); unit: years] — Caregivers were asked to estimate the number of years accompanying the enrolled patient to primary care doctor visits. Population: Caregivers only
  years
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 8.3 (9.4) | 8.9 (9.0) | 8.6 (9.2)
Caregiver - Symptoms of caregiving burden [Mean (Standard Deviation); unit: score on a scale] — Caregiver burden measured with 13-item Zarit Burden Inventory +1 global item as reported. Each item is scored 0-4 for a range of 0-52,higher scores indicating greater burden. Population: Caregivers only
  score on a scale
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 15.1 (10.2) | 14.6 (8.4) | 14.9 (9.4)
Caregiver - Symptoms of anxiety [Mean (Standard Deviation); unit: score on a scale] — Caregiver anxiety was measured using the Generalized Anxiety Disorder (GAD-7) which is a 7-item validated instrument that ask about symptoms of anxiety using a two-week recall period with response categories that vary from 0 ("not at all") to 3 ("nearly every day"). Item responses are summed to construct composite scores; range 0-21. Higher scores indicates more symptoms of anxiety. Population: Caregivers only
  score on a scale
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 3.4 (4.0) | 2.6 (2.9) | 3.0 (3.5)
Caregiver - Shared decision-making [Mean (Standard Deviation); unit: score on a scale] — Caregivers were asked to reflect on their interactions with the enrolled patient's primary care doctor and their team in the past 6 months using the CollaboRATE-10 scale. CollaboRATE-10 is a 3-item measure of the shared-decision making process on a 10-point anchored scale, ranging from 0 (no effort was made) to 10 (every effort was made). Participant's scores were summed and multiplied by 3.704 to transform the CollaboRATE-10 scale to 0 to 100. Higher scores indicate better interactions on shared-decision making process between caregiver and patient's primary care doctor. Population: Caregivers only
  score on a scale
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 84.8 (23.2) | 82.9 (23.1) | 83.9 (23.1)
Caregiver - Therapeutic Alliance [Mean (Standard Deviation); unit: score on a scale] — Caregivers were asked to reflect on the extent to which they felt a sense of mutual understanding, caring and trust with the enrolled patient's doctor. The 16-item Human Connection Scale (THC) was used to assess therapeutic alliance between patient and physician on a 4-point Likert scale ranging from 1-4 with various response categories depending on the relevance to question. The individual scores were summed; score range from 16-64. Higher scores indicate better sense of mutual understanding, caring and trust with patient's doctor. Population: Caregivers only
  score on a scale
    number analyzed (Participants) | 145 | 128 | 273
    (all) | 55.3 (9.4) | 53.3 (10.5) | 54.3 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Average Scores for Patient and Caregiver-Reported Quality of Communication at 6-Months
Description: The primary outcome assesses family-reported quality of communication with the primary care team using the 7-item end-of-life subscale of the validated Quality of Communication Scale. The scale for each item is from 0 ('Worst you can imagine') to 10 ('Best you can imagine'), with a range of 0-70 with higher scores indicating higher perceived quality of communication.
Time Frame: 6 months
Population: 216 represents the total number participants (patients, caregivers) assessed in the intervention group for this outcome at 6 months, and 194 represents the total number of participants (patients, caregivers) assessed in the control group for this outcome at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE | Minimally Enhanced Usual Care
Number analyzed (Participants) | 216 | 194
score on a scale
  Caregivers: number analyzed (Participants) | 108 | 97
  Caregivers | 3.41 (2.4) | 3.09 (2.4)
  Patients: number analyzed (Participants) | 108 | 97
  Patients | 3.06 (2.8) | 1.93 (1.9)

2. Secondary Outcome: Average Scores for Patient and Caregiver-Reported Readiness to Engage in Advance Care Planning at 6-months
Description: The Advance Care Planning Engagement Survey is a validated patient-reported questionnaire that assesses advance care planning process measures on a 5-point Likert scale. The outcome assesses a 6-item subscale of the Advance Care Planning Engagement Survey that includes parallel items for patient and family participants. The scale for each item is from 1 ("I have never thought about it") to 5 ("I have already done it"), with a range of 6-30 with higher scores indicating higher perceived readiness to engage in advance care planning.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHARE Group: The SHARE intervention group received a packet from the primary care practice including a person-family agenda setting checklist, blank advance directive, guide for communication with clinicians, instructions for completing proxy registration for the patient portal and an invitation to a facilitator led ACP conversation.
- Control Group: The control group received minimally enhanced usual care encompassing an introductory letter, the guide for communicating with clinicians and blank advance directive.
Arm/Group | SHARE Group | Control Group
Number analyzed (Participants) | 216 | 194
score on a scale
  Caregivers: number analyzed (Participants) | 108 | 97
  Caregivers | 27.01 (4.2) | 24.82 (6.9)
  Patients: number analyzed (Participants) | 108 | 97
  Patients | 17.25 (3.5) | 16.21 (4.6)

3. Secondary Outcome: Proportion of Patients With Documentation of Advance Directive Completion in the Electronic Health Record at 6-months
Description: Documentation of advance directive completion in the electronic health record is defined as having a durable power of attorney or a living will documented in the primary care electronic health record. The Medical Order for Life Sustaining Treatment (MOLST) will not be included for this outcome as the completion of a Maryland MOLST is mandatory in certain situations, such as on transfer between settings of care, and is not indicative of having had an advance care planning discussion or naming a durable power of attorney.
Time Frame: 6 months
Population: Data was not collected.
Arm/Group | SHARE | Minimally Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Average Scores for Bereaved Family-Reported Decisional Conflict
Description: Caregivers of patients who die are asked to assess their Decisional Conflict 2-3 months after patient's death. The Decisional Conflict Scale is a 16-item instrument scored on a 5-point Likert scale ranging from 0 ("strongly agree") to 4 ("strongly disagree").The 16 items are summed, divided by 16, then multiplied by 25 to yield scores that range from 0 (no decisional conflict) to 100 (extremely high decisional conflict). Higher scores indicate higher decisional conflict.
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Average Scores for Bereaved Family-Reported Decisional Regret
Description: Caregivers of patients who die are asked to assess their Decisional Regret 2-3 months after patient's death. This outcome assesses bereaved family-reported decisional regret using a 5-item instrument that assesses the extent to which decision-makers experience regret about care. Response options are assessed using a 5-item Likert scale in which scores of 1 indicate the least regret and 5 the most regret. Scores are then reduced by 1 point and multiplied by 25 for a scale that ranges in value from 0 to 100. Prior studies have categorized scores of 0 as no regret, 1 to 25 as mild regret, and more than 25 as heightened regret. Higher scores indicate stronger feelings of regret.
Time Frame: 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Average Scores for Bereaved Family Symptoms of Anxiety
Description: Caregivers of patients who die are asked to respond to questions about Symptoms of Anxiety 2-3 months after patient's death. This outcome assesses bereaved family symptoms of anxiety using the Generalized Anxiety Disorder 7-item questionnaire (GAD-7). The GAD-7 is a validated instrument that asks about symptoms of anxiety using a two-week recall period with response categories that vary from 0 ("not at all") to 3 ("nearly every day"). Item responses are summed to construct composite scores. Higher scores indicate more symptoms of anxiety.
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Average Scores for Bereaved Family-Reported Satisfaction With Care at the End-of-Life in Dementia
Description: Caregivers of patients who die are asked to assess their Satisfaction with Care at the End-of-life in Dementia 2-3 months after patient's death using the Satisfaction with Care at the End-of-Life in Dementia (SWC-EOLD). This is a 10-item instrument measured on a 4-point Likert scale that ranges from 1 ("strongly disagree") to 4 ("strongly agree") with a summary score ranging from 10-40 in which higher values indicate higher satisfaction. Higher scores indicate better satisfaction with care at the end-of-life in dementia.
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Patients Who Received Burdensome Care
Description: For patients who die while enrolled in the study by 24 months, this outcome assesses the proportion of patients who received burdensome care near the end of life. Burdensome care is defined as any intensive care unit use or life prolonging care (cardiopulmonary resuscitation, mechanical ventilation, tracheostomy, dialysis, artificial nutrition, chemotherapy) within 30 days of death using dates and services abstracted from medical records and the Chesapeake Regional Information System (CRISP), Maryland's Health Information Exchange, which includes all hospital encounters.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- SHARE Group: Patients; SHARE Group: Caregivers: The SHARE intervention group received a packet from the primary care practice including a person-family agenda setting checklist, blank advance directive, guide for communication with clinicians, instructions for completing proxy registration for the patient portal and an invitation to a facilitator led ACP conversation.
- Control Group: Patients; Control Group: Caregivers: The control group received minimally enhanced usual care encompassing an introductory letter, the guide for communicating with clinicians and blank advance directive.
Arm/Group | SHARE Group: Patients | Control Group: Patients | SHARE Group: Caregivers | Control Group: Caregivers
All-Cause Mortality (participants affected / at risk) | 34/145 | 29/128 | 0/145 | 2/128
Serious Adverse Events (participants affected / at risk) | 8/145 | 3/128 | 1/145 | 0/128
Other Adverse Events (participants affected / at risk) | 0/145 | 0/128 | 0/145 | 0/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SHARE Group: Patients (N=145) | Control Group: Patients (N=128) | SHARE Group: Caregivers (N=145) | Control Group: Caregivers (N=128)
Patient Hospitalized, Rehabilitated or Placed in Hospice (General disorders) | 8 | 3 | 1 | 0 — Caregivers reported to staff members during outreach for follow-up if patient was hospitalized, rehabilitated or placed in hospice. Patients

LIMITATIONS AND CAVEATS:
Primary care practices in one geographic location inhibits generalizability. Study is subject to Methodological challenges in the field, like including a lack of established and reliable gold standard measures of clinically meaningful endpoints.

Fielding quality of communication instrument has not been used primary care context to cognitively impairment patients and their care partners.

Observed treatment effects were variable by outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04593472/Prot_SAP_000.pdf